CLINICAL TRIAL: NCT02079870
Title: A Single-centre, Randomised, Double-blind Two-period Cross-over Trial Investigating the Effect of Semaglutide on Energy Intake, Appetite Sensations, Postprandial Glucose and Triglyceride Metabolism and Gastric Emptying in Obese Subjects Compared With Placebo
Brief Title: Trial Investigating the Effect of Semaglutide on Energy Intake, Appetite Sensations, Postprandial Glucose and Triglyceride Metabolism and Gastric Emptying in Obese Subjects Compared With Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3685; 2013-000012-24 (EudraCT Number); U1111-1138-2039 (Other: WHO)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Diabetes; Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Nutrition Disorders; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sema (Experimental): Two 12-week treatment periods separated by a wash-out period of 5-7 weeks. Finally, a follow-up visit is performed 5-7 weeks after last dosing
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Solution for subcutaneous (s.c. - under the skin) injection. 0.25 mg semaglutide once weekly for four weeks, 0.5 mg semaglutide once weekly for four weeks followed by 1.0 mg semaglutide once weekly for five weeks
  Arms: Sema
Drug: placebo — Solution for subcutaneous (s.c. - under the skin) injection
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the effect of semaglutide on energy intake, appetite sensations, postprandial glucose and triglyceride metabolism and gastric emptying in obese subjects compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent
* HbA1c (glycosylated haemoglobin A1c) below 6.5%
* A BMI (body mass index) between 30-45 kg/m^2 (both inclusive)

Exclusion Criteria:

* Females who are pregnant, breast-feeding or intend to become pregnant or is of childbearing potential and not using adequate contraceptive method (adequate contraceptive measures as required by local law or practice, UK requirements: adequate contraceptive measures are defined as established use of oral, injected or implanted hormonal methods of contraception, sterilisation, intrauterine device or intrauterine system, or consistent use of barrier methods together with the use of spermicide, and sexual abstinence)
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* Diagnosis of type 1 or 2 diabetes mellitus
* Anticipated change in lifestyle (e.g. eating, exercise or sleeping pattern) during the trial
* Use of any prescription or non-prescription medication which could interfere with trial pharmacokinetic or pharmacodynamic results, as judged by the investigator or specifically: 1) within 12 months prior to screening any weight lowering pharmacotherapy or pharmacotherapy that may cause weight gain, including systemic corticosteroids (except for a short course of treatment, i.e., 7-10 days), tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers, 2) within 3 months prior to screening use of statins, antihyperlipidemics including fibrates or nicotinic acid and its derivates, 3) supplementation with omega 3 fatty acids from 1 month prior to screening, 4) co-treatment with antihypertensive drugs is allowed if treatment has been stable for at least 1 month prior to screening and treatment should be kept unchanged during the trial
* Significant history of alcoholism or drug/chemical abuse within 1 year from screening, or a positive result of the urine drug screen or alcohol breath test, or consuming more than 21 units of alcohol per week for females and 28 units of alcohol per week for males (1 unit of alcohol equals ½ pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits)
* Smoking or use of any nicotine products (including nicotine patches, gum etc.) in the last 3 months prior to screening or a positive cotinine test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-07 (Actual)

PRIMARY OUTCOMES:
Ad libitum energy intake during a lunch meal (following a standardised breakfast meal) | After 12 weeks of treatment

SECONDARY OUTCOMES:
Mean postprandial increase (iAUC30-300min/270 min) in rating of overall appetite score (OAS) using Visual Analogue Scales (VAS) before and up to 300 minutes after intake of a standardised breakfast meal | After 12 weeks of treatment during a standardised meal test day
Incremental area under the 0-300 minutes glucose profile (iAUC0-300min,Glucose) following intake of a standardised breakfast meal | After 12 weeks of treatment during a standardised meal test day
Gastric emptying measured by the area under the 0-300 minutes plasma paracetamol concentration curve (AUC0-300min,para) following intake of a standardised breakfast meal (including 1500 mg paracetamol) | After 12 weeks of treatment during a standardised meal test day
Incremental area under the 0-480 minutes triglyceride profile (iAUC0-480min,TG) following intake of a standardised fat-rich meal | After 12 weeks of treatment during a standardised meal test day
Incidence of adverse events | From baseline to follow-up (5-7 weeks after last trial drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Leeds, United Kingdom

REFERENCES:
- [Result] Blundell J, Finlayson G, Axelsen M, Flint A, Gibbons C, Kvist T, Hjerpsted JB. Effects of once-weekly semaglutide on appetite, energy intake, control of eating, food preference and body weight in subjects with obesity. Diabetes Obes Metab. 2017 Sep;19(9):1242-1251. doi: 10.1111/dom.12932. Epub 2017 May 5. PMID 28266779
- [Result] Hjerpsted JB, Flint A, Brooks A, Axelsen MB, Kvist T, Blundell J. Semaglutide improves postprandial glucose and lipid metabolism, and delays first-hour gastric emptying in subjects with obesity. Diabetes Obes Metab. 2018 Mar;20(3):610-619. doi: 10.1111/dom.13120. Epub 2017 Oct 27. PMID 28941314
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com